CLINICAL TRIAL: NCT02877472
Title: Porous Tantalum Rods Improve the Hip Joint Function of Patients With Avascular Necrosis of the Femoral Head After Femoral Neck Fracture Surgery: a Randomized Controlled Trial
Brief Title: Porous Tantalum Rods Improve the Hip Joint Function of Patients With Avascular Necrosis of the Femoral Head
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qinghai University (Other)
Responsible Party: Principal Investigator, Heling Zhang, Attending Physician, Qinghai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QinghaiUH_003
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Femoral Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Patients with avascular necrosis of the femoral head after femoral neck fracture surgery will undergo core decompression and porous tantalum rod implantation (experimental group).
  Interventions: Device: porous tantalum rod
- Control group (Experimental): Patients with avascular necrosis of the femoral head after femoral neck fracture surgery will undergo core decompression (control group).
  Interventions: Procedure: core decompression

INTERVENTIONS:
Device: porous tantalum rod — Patients with avascular necrosis of the femoral head after femoral head fracture surgery receive treatment of core decompression and porous tantalum rod implantation
  Other Names: Experimental group
  Arms: Experimental group
Procedure: core decompression — Patients with avascular necrosis of the femoral head after femoral head fracture surgery will undergo core decompression.
  Other Names: Control group
  Arms: Control group

SUMMARY:
To confirm 1) whether, compared with core decompression alone, core decompression with porous tantalum rod implantation improves the hip joint function of patients with avascular necrosis of the femoral head after femoral neck fracture surgery, 2) whether porous tantalum rod shows favorable biocompatibility with the human body, and 3) whether this treatment method is feasible for treating avascular necrosis of the femoral head after femoral neck fracture surgery.

DETAILED DESCRIPTION:
History and current status of related studies: Femoral neck fracture can render the blood supply to the femoral head insufficient, leading to avascular necrosis of the femoral head. This often increases treatment difficulty and can have a strong influence on the recovery of hip joint function. Although core decompression for treatment of avascular necrosis of the femoral head has been largely used in clinical settings, the mid-term therapeutic effects are not satisfactory in some patients.

Biocompatibility is defined as the ability of a biomaterial, prosthesis, or medical device to perform with an appropriate host response. The biocompatibility of a bone implant and host influences the therapeutic effects. Therefore, biomaterials that are less likely to induce negative host responses may increase the therapeutic effects of such treatments for orthopedic diseases. A porous tantalum rod is a bone trabecula-like metal implant that is used to support weight-bearing areas of necrotic bone, preventing further collapse of the necrotic area. This implant has exhibited favorable effects in the early treatment of avascular necrosis of the femoral head. Although previous reports have focused on porous tantalum rod implantation for clinical treatment of avascular necrosis of the femoral head after fermoral neck fracture, few have assessed the long-term therapeutic effects or biocompatibility of porous tantalum rods.

Adverse events Possible adverse events include any expected or unexpected symptoms. If severe adverse events occur, information including the date of occurrence and measures taken related to the treatment of the adverse events will be reported to the principal investigator and the institutional review board within 24 hours.

Data collection, management, analysis, and open access Data collection: Case report forms with demographic data, disease diagnosis, accompanying diseases, drug allergy history, and adverse events will be collected , processed using Epidata software, collated, and then electrically recorded using a double-data entry strategy by data managers.

Data management: The locked electronic database will not be altered in any way, and will only be available to the project manager. Paper and electronic data regarding screening, informed consent, and clinical outcomes will be preserved at the Affiliated Hospital of Nantong University, China.

Data analysis: The electronic database will be made available to a professional statistician for statistical analysis. An outcome analysis report will be made by the statistician and submitted to the lead researchers. An independent data monitoring committee will supervise and manage the trial data with the goal of ensuring a scientific and stringent trial process, resulting in accurate and complete data.

Data open access: Anonymized trial data will be published at http://www.figshare.com.

Statistical analysis Statistical analysis will be performed by a statistician using SPSS 19.0 software and will follow the intention-to-treat principle. Normally distributed measurement data will be expressed as a mean, standard deviation, min, and max. Non-normally distributed measurement data will be expressed as a lower quartile (q1), median, and upper quartile (q3). McNemar's test will be used to compare the percentage of patients with excellent hip joint function as per Harris hip scores 12 months after surgery, the percentage of patients presenting with femoral head collapse, prosthesis loosening, peri-prosthesis infection, and incidence of complications 6 and 12 months after surgery. The Mann-Whitney U test will be used to compare the VAS score prior to and 1, 6, and 12 months after surgery. Statistical significance will be accepted when α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fracture nonunion as indicated by a clear fracture line 12 months after femoral neck fracture; avascular necrosis of the femoral head as shown by cystic degeneration, sclerosis, and uneven density on X-ray images and CT scans
* Patients with avascular necrosis of the femoral head after femoral neck fracture surgery who underwent internal fixation between 1 January 2016 and 31 May 2017
* Age 18-80 years
* Any sex and nationality
* Provision of signed informed consent to participate in the trial

Exclusion Criteria:

* Poor general health
* Chronic disease or history of surgery
* Alcohol abuse or long-term use of hormone drugs
* Unable or declines to cooperate with treatment and examination because of language and/or mental disorders
* Unable or declines to cooperate with rehabilitation treatment because of mental and/or psychological disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-10 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Harris hip scores | 12 months after surgery
  To evaluate the recovery of hip joint function. The Harris hip score ranges from 0-100 points with higher scores indicating better hip joint function. Hip joint function is scored as follows: ≥ 90 is excellent, 80-89 very good, 70-79 good, and < 70 poor.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | prior to and 1, 6, and 12 months after surgery
  To evaluate the severity of pain and ranges from 0-10, with higher scores indicating more severe pain.
Incidences of complications | 6 and 12 months after surgery
  To evaluate the safety of various implantation methods.

CONTACTS AND LOCATIONS:
Overall Officials: Heling Zhang, Master, Principal Investigator — Affiliated Hospital of Qinghai University
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China

IPD SHARING:
Plan to Share IPD: Undecided